CLINICAL TRIAL: NCT02050412
Title: A Pilot Study for the Determination of Allergenicity of Cat Dander Samples Obtained by Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Kuendig (Other)
Responsible Party: Sponsor-Investigator, Thomas Kuendig, PD Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZU-Scratch-Cat-001
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Cat Dander Allergy

ARMS (1):
- Cat fur scratch test (Other)
  Interventions: Other: Cat fur scratch test

INTERVENTIONS:
Other: Cat fur scratch test

SUMMARY:
Measurement of skin reactivity of cat dander samples obtained by different methods.

Subjects will be assessed for the study by of a conventional skin prick test with a positive (histamine), a positive (standardized cat dander extract) and a negative allergen control (a diluent) if they fulfil all other in- and exclusion criteria, too.

A screening prick test will be performed in order to confirm positivity (cat dander allergy).

A scratch test will be performed in participants after a positive screening prick test, in order to measure skin reactivity to cat dander, originating of three different body areas of the cat. For this purpose, a small amount of cat fur in solution with distilled water will be placed onto the volar aspect of both forearms after the skin has been scratched with a scratch lancet. The distilled water in which the cat hair was solved before will serve as negative control.

This procedure will be repeated with fur of the three different areas of the cat, always using triplicates (nine samples per cat).

From each of the 20 cats, nine samples will be tested on 20 subjects (one cat/subject).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female between 18 years to 65 years
* A positive clinical history with inhalant allergy presumably due to cat allergen.
* Positive screening prick test (mean wheal diameter ≥ 3 mm) when tested with already standardized cat allergen extract.
* Positive screening prick test (wheal diameter ≥ 3mm) to Histamine dihydrochloride 10mg/ml.

Exclusion Criteria:

* Impaired in understanding the nature, meaning and scope of the study or incapable of giving written informed consent,
* Participation in another clinical trial within the last 30 days and during the present study,
* Pregnant or lactating women,
* Positive skin reaction in the screening prick test to negative control,
* Currently suffering from allergy symptoms,
* History of systemic reactions to allergens,
* Severe diseases influencing the results of the present study by discretion of the investigator,
* Immunotherapy with the allergen preparation during the past two years,
* Skin lesions and excessive hair-growth in the skin test areas,
* Treatment with prohibited concomitant medications according to section 9.3 (protocol) with the exception of medications with local effects which will not influence the results of the skin tests,
* Alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary variable will be the wheal size area of the immediate phase reaction in mm² | measured after 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, University Hospital and University Zurich, Zurich, Canton of Zurich, Switzerland